CLINICAL TRIAL: NCT05286645
Title: Intervention Effect of High Definition Transcranial Direct Current Stimulation (HD-tDCS) on Depressive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, WANG KAI, Director of medical psychological department, Anhui Medical University, Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AHMU-tdcs-depression
Record Dates: First submitted 2022-01-13; First posted 2022-03-18 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2024-09

CONDITIONS: Transcranial Direct Current Stimulation; Functional Magnetic Resonance Imaging; Depressive Disorder
Keywords: Transcranial Direct Current Stimulation; Functional Magnetic Resonance Imagin; Depressive Disorder
MeSH Terms: conditions — Depressive Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real stimulation (Active Comparator): Participants will receive active tDCS once daily for two weeks. The anode was placed over Fz with return electrodes placed at Fpz, Cz, F3 and F4. Fourteen 2-mA sessions (ramp-up and ramp-down periods of 30 and 30 seconds, respectively) were applied for 20 minutes each day over 14 consecutive sessions.
  Interventions: Device: High definition transcranial direct current stimulation
- sham stimulation (Placebo Comparator): Participants will receive sham tDCS once daily for two weeks. Sham HD-tDCS was delivered using the same protocol and current intensity, but the period of active stimulation was only during the ramp-up and ramp-down periods of 30 and 30 seconds.
  Interventions: Device: sham high definition transcranial direct current stimulation

INTERVENTIONS:
Device: High definition transcranial direct current stimulation — tDCS is described as a non-invasive form of brain stimulation that uses a low-intensity, constant current applied directly to the head through scalp electrodes.
  Arms: real stimulation
Device: sham high definition transcranial direct current stimulation — Sham HD-tDCS was delivered using the same protocol and current intensity, but the period of active stimulation was only during the ramp-up and ramp-down periods of 30 and 30 seconds.
  Arms: sham stimulation

SUMMARY:
To investigate the intervention effect of high definition transcranial direct current stimulation (HD-tDCS) on somatic symptoms in patients with depressive disorder and its underlying neural mechanism by MRI.

DETAILED DESCRIPTION:
Depressive disorder is a major public health and safety problem around the world. Patients with depression often performe symptoms such as anhedonia, lack of motivation, somatic symptoms, and even suicidal ideation and behavior. The purpose of this study was to study the relieving effect of high definition transcranial direct current stimulation (HD-tDCS) on the symptoms of depression.

60 patients with depressive disorder diagnosed by DSM-5 were recruited from the fourth people's Hospital of Hefei and the first affiliated Hospital of Anhui Medical University. All participants underwent a structured interview and routine laboratory examination before and after receiving HD-tDCS. After meeting the inclusion criteria and obtaining informed consent. Each participant will complete the clinical evaluation, functional magnetic resonance imaging (fMRI) and HD-tDCS treatment conducted by trained researchers at the Neuropsychological Synergetic Innovation Center of Anhui Medical University. All the participants were randomized (1:1) to receive "active" or "sham" treatment protocol. The anode was placed over Fz with return electrodes placed at Fpz, Cz, F3 and F4. Fourteen 2-mA sessions (ramp-up and ramp-down periods of 30 and 30 seconds, respectively) were applied for 20 minutes each day over 14 consecutive sessions. Sham HD-tDCS was delivered using the same protocol and current intensity, but the period of active stimulation was only during the ramp-up and ramp-down periods of 30 and 30 seconds.

Before and after the HD-tDCS treatment, the patients had receiving a battery measure of neuropsychological tests and Magnetic resonance imaging scan in multimodalities. Neuropsychological assessment included MoCA, Stroop Test, VFT, DST, AVLT, HAMD, HAMA, PHQ15, BSS(Beck scale for suicide ideation),ISI,SDS, RRS, TEPS, AES, FPQ, PVAQ and AAS. Multimodal fMRI includes 3D-T1, rs-fMRI, DTI and ASL.

Neuropsychological evaluation and magnetic resonance imaging data were obtained again 24 hours after the last treatment. The symptoms of the patients were followed up one month after the end of treatment.They were instructed to focus their answers on the past week. Afterwards, they were unblinded by the study coordinator.

ELIGIBILITY:
Inclusion Criteria:

* the patients were diagnosed by more than 2 psychiatrists and met the diagnostic criteria of DSM-5 for depression, and HAMD>17, PHQ-15>5.
* the age ranged from 18 to 60 years old
* right-handed
* stable dose of medication for at least 4 weeks or no history of antidepressive drugs before intervention

Exclusion Criteria:

* accompanied by severe somatic diseases, such as severe heart, liver, renal insufficiency and so on.
* accompanied by other neurological diseases, such as stroke, epilepsy and so on.
* accompanied by other mental disorders, such as drug abuse, schizophrenia, schizophrenic affective disorder, hysteria, autism and so on.
* patients with MRI taboos or factors affecting imaging quality, such as cardiac pacemaker, cochlear implant, cardio-cerebrovascular metal stent, metal denture, etc.
* pregnancy and breastfeeding.
* previous physical treatment (electroconvulsive therapy or tDCS).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 57 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
the change of somatic symptoms in active group and sham group at post-treatment and follow-up visit. | Baseline, Week 2 and Week 8.
  the somatic symptoms were assessed by PHQ-15 scale.
the percentage decrease in PHQ-15 scores in active group and sham group at post-treatment and follow-up visit. | Baseline, Week 2 and Week 8.
  The percentage of decrease in scores was measured using the following formula: (pretreatment scores - post-treatment scores)/pretreatment scores × 100 %).
the number of somatic responders in active group and sham group at post-treatment and follow-up visit. | Baseline, Week 2 and Week 8.
  Responders were defined as patients who had a ≥ 50% decrease in the PHQ-15 score.

SECONDARY OUTCOMES:
the change of depressive symptoms in active group and sham group at post-treatment and follow-up visit. | Baseline, Week 2 and Week 8.
  the depressive symptoms were assessed by HAMD scale.
the percentage decrease in HAMD scores in active group and sham group at post-treatment and follow-up visit. | Baseline, Week 2 and Week 8.
  The percentage of decrease in scores was measured using the following formula: (pretreatment scores - post-treatment scores)/pretreatment scores × 100 %).
the number of depressive responders in active group and sham group at post-treatment and follow-up visit. | Baseline, Week 2 and Week 8.
  Responders were defined as patients who had a ≥ 50% decrease in the HAMD score.

CONTACTS AND LOCATIONS:
Overall Officials: Ting Zhang, Study Chair — Anhui Medical University
Locations (1):
- Anhui Medical University, Hefei, China

DOCUMENTS (1):
  • Study Protocol (2025-12-25): https://cdn.clinicaltrials.gov/large-docs/45/NCT05286645/Prot_000.pdf